CLINICAL TRIAL: NCT01684631
Title: Prospective, Multicentric, Observational Cohort Study for the Evaluation of Implant Survival in Patients With a Metal-on-Metal Pinnacle(R) Ultamet(TM) Device in Conventional Total Hip Joint Replacement.
Brief Title: Evaluation of Implant Survival in Patients With a Pinnacle Ultamet Device in Conventional Total Hip Joint Replacement
Status: Completed | Type: Observational
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Other Study IDs: 27062008
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Arthropathy of Hip
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hip arthroplasty: Patients implanted with a PINNACLE® ULTAMET™ Metal-on-Metal implant for conventional total hip arthroplasty for the treatment of a severe hip disease or true femoral cervical fracture.
  Interventions: Device: Total Hip arthroplasty

INTERVENTIONS:
Device: Total Hip arthroplasty

SUMMARY:
The objective is to evaluate the implant survival rate for patients implanted with a PINNACLE® ULTAMET™ Metal-on-Metal implant for conventional total hip arthroplasty for the treatment of a severe hip disease and true femoral cervical fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients susceptible to receive a PINNACLE® ULTAMET™ implant as per routine practice

Exclusion Criteria:

* Patient refusal to participate to the data collection
* Pregnant woman
* Patients age is less than 18 years old
* The planned intervention is a revision of a previous intervention on the studied hip joint
* Previous metal implant, except for pure titanium or titanium alloys
* Exposure to cobalt and chromium that could influence serum metal ions levels
* Planned bilateral intervention
* Patient residing outside France
* Patient not implanted with a Pinnacle(R) ULTAMET(TM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients susceptible to receive a PINNACLE® ULTAMET™ implant
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2009-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Implant Survival Rate | up to 5 years
  Implant Survival Rate as the duration of PINNACLE® ULTAMET™ implantation for the follow-up duration, free of revision surgery, whatever the cause.

SECONDARY OUTCOMES:
Harris Hip Score | pre-operative, 1, 2, 3, 5 years
  Measure of hip function using the Harris Hip Score

OTHER OUTCOMES:
Cobalt and Chromium serum concentration | 3 to 6 Months, 1, 2, 3, 5 years
  Descriptive analysis of patient serum concentration of Cobalt and Chromium
Adverse Event Frequency | Per-operative, 3 to 6 Months, 1, 2, 3, 5 years
  Descriptive Analysis of Adverse Event Frequency for the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Toupin, MD, Principal Investigator — Clinique Saint Hilaire Rouen, France 76000
Locations (6):
- France (6):
  - Clinique Herbert, Aix-les-Bains
  - Clinique Bonnefon, Alès
  - Centre Hospitalier Georges Renon, Niort
  - Clinique Saint Hilaire, Rouen
  - Clinique Pasteur, Royan
  - Clinique Mutualiste Saint Etienne, Saint-Etienne

REFERENCES:
- [Background] Harris WH. Traumatic arthritis of the hip after dislocation and acetabular fractures: treatment by mold arthroplasty. An end-result study using a new method of result evaluation. J Bone Joint Surg Am. 1969 Jun;51(4):737-55. No abstract available. PMID 5783851